CLINICAL TRIAL: NCT02593968
Title: a Multi-sites, Randomized, Parallel, Placebo-Controlled Clinical, Pilot Study to Evaluated the Efficacy and Safety of Recombinant Human Interferon Alpha-2b Gel (Yallaferon®) in HPV Infection
Brief Title: Yallaferon in Chinese Population
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zhaoke-1504-Yallaferon
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): subject were treated 3 periods with Yallaferon®; each period has interval 10 days ; one period included Yallaferon application for every other day for 10 times
  Interventions: Drug: Recombinant Human Interferon a-2b Gel
- Plcaebo (Placebo Comparator): subject were treated 3 periods with Yallaferon® Plcaebo; each period has interval 10 days; one period included Yallaferon application for every other day for 10 times
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant Human Interferon a-2b Gel
  Arms: Treatment
Drug: Placebo
  Arms: Plcaebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Yallaferon in Chinese population with HPV-16 and/or HPV-18.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 65 years of age the sex life of female patients;
* High-risk HPV 16 and/or 18 positive
* Agree to sign ICF

Exclusion Criteria:

* Cervical intraepithelial neoplasia (CIN);
* Combined with a severe fungal, trichomonas vaginitis;
* Severe primary diseases associated with cardiovascular, liver, kidney and hematopoietic system;
* Allergies or allergy to the drug known ingredients.
* Within 30 days to accept other clinical trials of drugs or are participating in clinical trials;
* Pregnant and lactating women and to be pregnant women;
* The researchers do not consider it appropriate clinical trials.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
HPV-16 and/or HPV-18 negative conversion rate | 3 months
  hr-HPV DNA negative conversion rate will be evaluated at 3 months after treatment in treatment and placebo group; calculation method: proportion of patient with HPV negative expression

SECONDARY OUTCOMES:
HPV-16 and/or HPV-18 negative conversion rate | 6 months
  hr-HPV DNA negative conversion rate will be evaluated at 6 months after treatment in treatment and placebo group; calculation method: proportion of patient with HPV negative expression
HPV-16 and/or HPV-18 negative conversion rate | 9 months
  hr-HPV DNA negative conversion rate will be evaluated at 9 months after treatment in treatment and placebo group; calculation method: proportion of patient with HPV negative expression
HPV-16 and/or HPV-18 negative conversion rate | 12 months
  hr-HPV DNA negative conversion rate will be evaluated at 12 months after treatment in treatment and placebo group; calculation method: proportion of patient with HPV negative expression
reinfection at 12 months | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China